CLINICAL TRIAL: NCT03487016
Title: A Multicenter Randomized Phase II Study to Determine the Optimal First-line Chemotherapy Regimen in Patients With Metastatic Pancreatic Cancer
Brief Title: First-line Therapy in Metastatic PDAC
Acronym: FOOTPATH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, PD Dr. med. Volker Heinemann, Professor of Medicine, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-003496-54
Record Dates: First submitted 2018-03-04; First posted 2018-04-03 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Pancreatic Cancer; First line; Metastatic
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Fluorouracil; irinotecan sucrosofate; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A: Gemcitabine/nab-Paclitaxel (Standard) (Active Comparator): Nab-paclitaxel 125 mg/m2, i.v. infusion over about 30 minutes followed by Gemcitabine 1000 mg/m2 as a 30-minute i.v. infusion on D1, D8, D15 of a 28-day cycle.
  Treatment is given until disease progression or the occurrence of unacceptable toxicity.
  Interventions: Drug: Gemcitabine; Drug: Nab-paclitaxel
- B: NAPOLI regimen (Experimental): On Day 1 of a 14-day cycle:
  Liposomal irinotecan 80 mg/m2 i.v. over about 90 minutes followed by Folinic acid 400 mg/m2 i.v. over about 30 minutes followed by 5-FU 2400 mg/m2 i.v. over about 46 h (pump)
  Treatment is given until disease progression or the occurrence of unacceptable toxicity.
  Interventions: Drug: 5-FU; Drug: Irinotecan Liposomal Injection
- C: seq-NAPOLI-FOLFOX (Experimental): The NAPOLI regimen and the mFOLFOX6 regimen are applied in an alternating fashion, starting with the NAPOLI regimen.
  NAPOLI:
  On Day 1 of a 14-day cycle:
  Liposomal irinotecan 80 mg/m2 i.v. over about 90 minutes followed by Folinic acid 400 mg/m2 i.v. over about 30 minutes followed by 5-FU 2400 mg/m2 i.v. over about 46 h (pump)
  mFOLFOX6:
  On Day 1 of a 14-day cycle:
  Oxaliplatin 85 mg/m2 as i.v. infusion over 2 to 6 hours according to local practice at trial site Folinic acid 400 mg/m2 as i.v. infusion; infusion duration according to local practice at trial site followed by 5-FU 2400 mg/m2 i.v. over about 46 h (pump)
  Treatment is given until disease progression or the occurrence of unacceptable toxicity.
  Interventions: Drug: 5-FU; Drug: Irinotecan Liposomal Injection; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Gemcitabine — Arm A
  Other Names: Gemzar
  Arms: A: Gemcitabine/nab-Paclitaxel (Standard)
Drug: Nab-paclitaxel — Arm A
  Other Names: Abraxane
  Arms: A: Gemcitabine/nab-Paclitaxel (Standard)
Drug: 5-FU — Arm B Arm C
  Other Names: 5-Fluoruracil
  Arms: B: NAPOLI regimen; C: seq-NAPOLI-FOLFOX
Drug: Irinotecan Liposomal Injection — Arm B Arm C
  Other Names: Onivyde
  Arms: B: NAPOLI regimen; C: seq-NAPOLI-FOLFOX
Drug: Oxaliplatin — Arm C
  Other Names: Trans-l-diaminocyclohexanoxalatoplatin
  Arms: C: seq-NAPOLI-FOLFOX

SUMMARY:
The overarching hypothesis of this trial is that the NAPOLI regimen and alternating cycles of NAPOLI and mFOLFOX6 (seq-NAPOLI-FOLFOX) are superior to the current standard of care gemcitabine/nab-paclitaxel. Furthermore, we propose that the NAPOLI regimen and seq-NAPOLI-FOLFOX display favourable safety profiles and allow for longer first line treatment and higher rate of transition into the second line setting.

DETAILED DESCRIPTION:
Pancreatic ductal adenocarcinoma (PDAC) remains an almost uniformly lethal disease. Although there has been significant progress in understanding of the underlying molecular biology of pancreatic cancer, this progress has not translated into substantially better outcome.

Alarmingly, the number of pancreatic cancer cases is constantly rising and pancreatic cancer will be the second most frequent cause of cancer related death by 2030.

Accordingly, novel therapeutic strategies for patients with pancreatic cancer are desperately needed.

Recently, the combination of gemcitabine and nab-paclitaxel proofed to be superior when compared to single agent gemcitabine (overall survival [OS] 8.7 months in the nab-paclitaxel/gemcitabine group versus 6.6 months in the gemcitabine group; hazard ratio for death, 0.72; 95% confidence interval [CI], 0.62 to 0.83; P<0.001). Consequently, this combination therapy is now regarded as a standard treatment option for patients with metastatic pancreatic cancer and should therefore serve as control for future clinical studies.

Furthermore, the combination of 5-fluorouracil (5-FU), irinotecan and oxaliplatin (FOLFIRINOX) was found to be more effective in the treatment of metastatic pancreatic cancer when compared to gemcitabine monotherapy (overall survival 11.1 month in the FOLFIRINOX group versus 6.8 months in the gemcitabine group - hazard ratio for death, 0.57; 95% confidence interval [CI], 0.45 to 0.73; P<0.001). However, this increased activity came at the cost of higher treatment-related side effects.

Recently, the NAPOLI-1 trial yielded promising results for the combination of liposomal irinotecan (nal-Iri) in combination with 5-FU/folinic acid (FA) in patients pretreated with a gemcitabine-based first-line regimen.

Finally, Phase II data show promising efficacy and favorable toxicity with conventional FOLFIRI.3 in the treatment of advanced pancreatic cancer.

Furthermore, studies in colorectal cancer demonstrated a comparable efficacy and favorable toxicity when comparing conventional FOLFOXIRI (+ bevacizumab) and sequential FOLFOXIRI (alternating FOLFOX and FOLFIRI) in combination with bevacizumab.

With these novel treatment options at hand it is imperative to define the optimal first-line treatment modality in order to allow for an optimized treatment sequence to ensure for maximal success with acceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years of age and ≤ 75 years
* Histologically (not cytologically) confirmed diagnosis of metastatic pancreatic ductal adenocarcinoma (PDAC) [Stage IV according to UICC TNM edition 8 of 201622: each T, each N, M1]
* No option for surgical resection or radiation in curative intent
* At least one unidimensionally measurable tumor lesion (according to RECIST 1.1)
* ECOG performance status 0 - 1
* Life expectancy at least 3 months
* Adequate hepatic, renal and bone marrow function, defined as:
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
* Haemoglobin ≥ 9 g/dL
* Thrombocytes ≥ 100 x 109/L
* Total bilirubin ≤ 1.5 x ULN. Patients with a biliary stent may be included provided that bilirubin level after stent insertion decreased to ≤ 1.5 x ULN and there is no cholangitis.
* AST/GOT and/or ALT/GPT ≤ 2.5 x ULN or in case of liver metastasis ≤ 5 x ULN)
* Serum creatinine within normal limits or creatinine clearance ≥ 60 mL/min/1.73 m2 as calculated by CKD-EPI formula for patients with serum creatinine levels above or below the institutional normal value.
* Females of childbearing potential (FCBP) must have a negative highly sensitive serum pregnancy test within 7 days of the first administration of study treatment and they must agree to undergo a further pregnancy tests at monthly intervals and at the end of treatment visit and FCBP must either agree to use and be able to take highly effective contraceptive birth control methods (Pearl Index < 1) during the course of the study and for at least 1 month after last administration of study treatment. Complete sexual abstinence is acceptable as a highly effective contraceptive method only if the subject is refraining from heterosexual intercourse during the entire study treatment and at least one month after the discontinuation of study treatment and the reliability of sexual abstinence is in line with the preferred and usual lifestyle of the subject. A female subject following menarche is considered to be of childbearing potential unless she is naturally amenorrhoeic for ≥ 1 year without an alternative medical reason, or unless she is permanently sterile.
* Males must agree to use condoms during the course of the trial and for at least 6 months after last administration of study drugs or practice complete abstinence from heterosexual intercourse.
* Signed and dated informed consent before the start of any specific protocol procedures
* Patient's legal capacity to consent to study participation

Exclusion Criteria:

* Locally advanced PDAC without metastasis
* Symptomatic/clinically significant ascites (expected indication for repeated paracentesis)
* Known metastatic disease to the brain. Brain imaging is required in symptomatic patients to rule out brain metastases, but is not required in asymptomatic patients.
* Previous palliative chemotherapy or other palliative systemic tumor therapy for metastatic disease of PDAC
* Previous gemcitabine or 5-FU based treatment with exception of gemcitabine/fluoropyrimidine based treatment applied in the neoadjuvant or adjuvant setting (before/after potential curative R0 or R1 resection) and if the neoadjuvant/adjuvant chemotherapy was terminated at least 6 months before randomization
* Previous radiotherapy of PDAC with exception of radiotherapy in the context of a neoadjuvant or adjuvant treatment setting that was terminated at least 6 months before randomization
* Any major surgery within the last 4 weeks before randomization
* Clinically significant decrease in performance status within 2 weeks of intended first administration of study medication (by medical history)
* Severe tumor-related cachexia and/or known weight loss > 15% within one month before study enrollment
* Pre-existing polyneuropathy ≥ grade 2 according to CTCAE version 4.03
* Gastrointestinal disorders that might interfere with the absorption of the study drug and gastrointestinal disorders with diarrhoea as a major symptom (e.g. Crohn's disease, malabsorption), and chronic diarrhoea of any aetiology CTCAE version 4.03 grade ≥ 2
* Any other severe concomitant disease or disorder, which could influence patient's ability to participate in the study and his/her safety during the study or interfere with interpretation of study results e.g. active infection, uncontrolled hypertension, clinically significant cardiovascular disease e.g. cerebrovascular accident (≤ 6 months before study start), myocardial infarction (≤ 6 months before study start), unstable angina, heart failure ≥ NYHA functional classification system grade 2, severe cardiac arrhythmia requiring medication, metabolic dysfunction, severe renal disorder.
* Any other malignancies than PDAC within the last 5 years before study start, except for adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer
* Hypersensitivity to the study drugs or to any of the excipients or to compounds with similar chemical or biologic composition
* Use of strong CYP3A4 inhibitors (CYP3A4 inhibitors have to be discontinued at least one week prior to start of study treatment).

Use or strong UGT1A1 inhibitors or strong CYP3A4 inducers unless there are no therapeutic alternatives.

* Known glucuronidation deficiency (Gilbert's syndrome) (specific screening not required)
* Known DPD deficiency (specific screening not required)
* Requirement for concomitant antiviral treatment with sorivudine or brivudine
* Continuing abuse of alcohol, drugs, or medical drugs
* Pregnant or breast-feeding females or FCBPs unable to either perform highly effective contraceptive measures or practice complete abstinence from heterosexual intercourse
* Current or recent (within 4 weeks prior to randomization) treatment with an investigational drug or participation in an investigational clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 60 months
  PFS

SECONDARY OUTCOMES:
Overall survival | 60 months
  OS
Objective response rate | 60 months
  ORR
Disease control rate | 60 months
  DCR
Duration of study treatment | 60 months
  Time on therapy
Type, incidence, causal relationship and severity of adverse events according to NCI CTCAE version 4.03 | 60 months
  Safety
Efficacy of second-line chemotherapy | 60 months
  Second Line Therapy I
  Assessed through progression free survival after initiation of second-line therapy.
Choice of second-line chemotherapy | 60 months
  Second Line Therapy II
  Type of second line therapy will be recorded in a descriptive manner based on available health records.
Duration of second-line chemotherapy | 60 months
  Second Line Therapy III
Quality of life as assessed by EORTC-QLQ-C30 | 60 months
  Quality of life will be assessed by the European Organisation for Research and Treatment of Cancer (EORTC) core Quality of Life Questionnaire (QLQ).
  The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale.
  All of the scales ands ingle-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
  Scoring is done based on the following document: EORTC QLQ-C30 Scoring Manual

OTHER OUTCOMES:
Molecular subtypes of pancreatic cancer as predictors of response to chemotherapy | 60 months
  Translational 1
Evaluation of radiologic early tumor shrinkage | 60 months
  ETS will be assessed after 8 weeks of treatment.
  Early tumour shrinkage (ETS) will be analysed based on sum of longest diameters of target lesions (SLD).
  Shrinkage will be classified as ETS (shrinkage by ≥20%), mETS (minor shrinkage by 0% - <20%), mPD (minor progression by >0% - <20%), PD (progression by ≥20% or new lesion).
  In all caculations, shrinkage will be expressed as a positive denominator.
Evaluation of radiologic depth of response | 60 months
  Radiologic depth of response is (DpR) is defined as the percentage of tumour shrinkage, based on sum of longest diameters of target lesions (SLD) observed at the lowest point (nadir) compared with baseline imaging.
  Tumour shrinkage (TS) will be classified as: (shrinkage by ≥20%), mTS (minor shrinkage by 0% - <20%), mPD (minor progression by >0% - <20%), PD (progression by ≥20% or new lesion).
  In all caculations, shrinkage will be expressed as a positive denominator.
Kinetics of circulating tumor DNA during first-line chemotherapy | 60 months
  Translational 1
  Circulating tumour DNA will be assessed through polymerase chain reaction based techniques and the concentration will be denominated as "ng/mL of plasma". Samples will be collected at the start of each cycle to allow for the detection of changing concentrations during first-line treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Volker Heinemann, MD, Principal Investigator — LMU Munich
Locations (1):
- Klinikum der Universitaet Muenchen - Campus Grosshadern, Munich, Germany